CLINICAL TRIAL: NCT03466658
Title: Preoperative Application of Low-level Microcurrent Dressing (Jumpstart) for Decolonization of P. Acnes Before Shoulder Surgery
Brief Title: Preoperative Jumpstart for Decolonization of P. Acnes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unexpected culture contamination potentially due to a testing error
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, H Mike Kim, MD, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00009349
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Shoulder Arthropathy Associated With Other Conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- JumpStart group (Experimental): This group will have the JumpStart dressing pre-operatively. Intervention: JumpStart dressing
  Interventions: Device: JumpStart Antimicrobial Wound Dressing
- Control group (No Intervention): This group will have no intervention pre-operatively. Intervention: none

INTERVENTIONS:
Device: JumpStart Antimicrobial Wound Dressing — A novel, wireless, low-level microcurrent-generating antimicrobial device (JumpStart) is a sterile single layer dressing consisting of a matrix of alternating silver (Ag) and zinc (Zn) dots that are held in positions on a polyester substrate with biocompatible binder. Dressing is then activated in the presence of a conductive fluid, which may come from wound exudate or exogenous fluids, such as saline. It has been observed, in vitro, to exhibit electricidal effect in the presence of antibiotic and multidrug resistant clinical wound isolates.
  Arms: JumpStart group

SUMMARY:
The objective of the study is to evaluate the efficacy of preoperative treatment with a novel, wireless, low-level microcurrent-generating antimicrobial device (brand name: JumpStart) in preventing the spread of Propionibacterium acnes in patients receiving open or arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
The spread of multi-drug resistant bacteria and financial burden of periprosthetic joint infection exacerbate the need for treatments to address pathogenic contamination and expedite healing. Although rare, these infections can place a great financial burden on the health care system and are often associated with increased hospital length of stay, compromised function, reduced quality of living, and increased likelihood of follow-up surgeries. Bacterial infection can further compound this problem with the widespread, prolonged use of prolonged antimicrobial prophylaxis. It is know that there is a high frequency of infections after open and arthroscopic shoulder surgery caused by Propionibacterium acnes. Because P. acnes normally colonizes under the epidermal layer in sebaceous glands, topical skin preparations, skin cleansers, and antibiotics may be unable to completely penetrate the deep layers of the skin to eradicate its colonization in all layers of the skin.

A novel, wireless, low-level microcurrent-generating antimicrobial device has been observed, in vitro, to exhibit electricidal effect in the presence of antibiotic and multidrug resistant clinical wound isolates. These energy-based systems were originally employed to augment wound healing process, reduce infection, and address edema and pain in the recent decades. Low-level microcurrents have been recently expanded into the orthopedic space as a bacterial growth inhibitor both in vitro and in vivo. Procellera (JumpStart) is a sterile single layer dressing consisting of a matrix of alternating silver (Ag) and zinc (Zn) dots that are held in positions on a polyester substrate with biocompatible binder. Dressing is then activated in the presence of a conductive fluid, which may come from wound exudate or exogenous fluids, such as saline.

Many studies have been done already on the wound healing and pain management properties of JumpStart, but only few have explored its bactericidal properties. To date, no MRSA strains have been found to possess Ag-resistant genes, and there is no known mechanism of bacterial resistance to all heavy metal ions. However, studies have suggested that the widespread and uncontrolled use of Ag+ in wound care may result in more bacteria developing resistance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Scheduled to receive open or arthroscopic shoulder surgery

Exclusion Criteria:

* 17 years old or younger
* Pregnant women
* Prisoners
* Non-English speaking or unable to understand consent
* History of any prior shoulder surgery
* History of previous shoulder infection or clinical signs of preoperative infection
* History of taking any antibiotic(s) within 4 weeks prior to the scheduled shoulder surgery
* Active acne or skin inflammatory disorders (psoriasis, eczema, etc) in the shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyunmin Kim, MD, Principal Investigator — Penn State Bone and Joint Institute
Locations (1):
- Penn State Bone and Joint Institute, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the Penn State Health Orthopedics Clinic for indications of open or arthroscopic shoulder surgery.
Pre-assignment Details: 17 participants met inclusion criteria and were enrolled. 3 participants withdrew prior to study intervention.
Units Other Than Participants: Shoulder
Groups:
- All Participants: Enrolled participants served as their own control. The surgical shoulder served as the Treatment Shoulder with the Jumpstart dressing intervention, while the normal non-operative contralateral shoulder served as the Control Shoulder.
Period: Overall Study
Arm/Group | All Participants
Started | 17; 34 Shoulder
Completed | 14; 28 Shoulder
Not Completed | 3; 6 Shoulder
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Enrolled participants served as their own control, where both shoulders of each participant will be included for the study. The surgical side shoulder will serve as a Treatment Shoulder with the Jumpstart dressing intervention, while the normal non-operative contralateral shoulder will serve as a Control Shoulder.
Arm/Group | All Participants
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 61 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Enrolled participants served as their own control, where both shoulders of each participant will be included for the study. The surgical side shoulder will serve as a Treatment Shoulder with the Jumpstart dressing intervention, while the normal non-operative contralateral shoulder will serve as a Control Shoulder.
  participants
    United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Presence of Propionibacterium Acnes in Skin Biopsies During Surgery
Description: The primary outcome measures the intraoperative culture results (e.g. positive vs negative, days to positive conversion) for P. acnes by evaluating bacterial cultures from punch skin biopsies at the time of the surgery.
Time Frame: 7 days post-biopsy
Population: Data not analyzed due to unexpected culture contamination.
Arm/Group | JumpStart Group | Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 7 days post shoulder surgery
Arm/Group | JumpStart Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT03466658/Prot_SAP_000.pdf